CLINICAL TRIAL: NCT06917573
Title: Phase II Clinical Trial With an Adaptive Design According to Response to Cemiplimab Monotherapy Using ctDNA and Subsequent Treatment With Chemotherapy (CT) and Cemiplimab or Cemiplimab Monotherapy in First Line Advanced NSCLC Patients
Brief Title: PALACE: Cemiplimab Trial According to ctDNA Levels
Acronym: PALACE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 22/01_PALACE; 2024-518812-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Lung Diseases; Stage IV Non-small Cell Lung Cancer; Stage III Non-small Cell Lung Cancer; Respiratory Tract Neoplasms; Thoracic Neoplasms
Keywords: Cemiplimab; ctDNA levels; Chemotherapy; Non-resectable non-small cell lung cancer
MeSH Terms: conditions — Lung Diseases; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms | interventions — cemiplimab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): A. Cemiplimab monotherapy
  - Cemiplimab
  Cemiplimab will be administered in monotherapy for 2 cycles. After 2 cycles of treatment and after response evaluation according to RECIST criteria and ctDNA quantification, patient will receive cemiplimab + chemotherapy or continue treatment with cemiplimab monotherapy
  Cemiplimab monotherapy will be administered until disease progression, unacceptable toxicity, loss of clinical benefit as judged by the investigator or up to a maximum of 2 years of treatment.
  B. Cemiplimab + chemotherapy
  The treatment with chemotherapy will be selected according to investigator's choice. Carboplatin and Pemetrexed or Carboplatin plus taxanes is recommended.
  Interventions: Drug: Cemiplimab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cemiplimab — Patients will receive Cemiplimab administered by IV infusion over 30 minutes every 28 days (Q3W) until disease progression, unacceptable toxicity, loss of clinical benefit as judged by the investigator or up to a maximum of 2 years of treatment.
  Structure: is a high affinity hinge-stabilized IgG4P human antibody to the PD-1receptor (PDCD1, CD279) that blocks PD 1/PD L1 mediated T cell inhibition. Binding of the PD-1 ligands PD-L1 and PD-L2, to the PD-1 receptor found on T cells, inhibits T-cell proliferation and cytokine production. Upregulation of PD-1 ligands occurs in some tumors and signaling through this pathway can contribute to inhibition of active T-cell immune surveillance of tumors.
  Route of administration: Intravenous infusion.
  Other Names: REGN2810
Drug: Carboplatin — Patients will receive Carboplatin administered by IV infusion for 2 cycles.
  Structure: The cis-diamino (cyclobutane-1, 1 dicarboxylate) platin.
  Stability: 24 hours at ambient temperature in 5% glucose, glucosaline or physiologic saline. It is recommended not to dilute with chlorinated solutions since this could affect the carboplatin.
  Route of administration: Intravenous infusion.
  Other Names: Paraplatin; Carboplatine
Drug: Paclitaxel — Patients will receive Paclitaxel administered by IV infusion for 2 cycles.
  Structure: A diterpene whose composition is: 5b, 20- epoxy-1, 2a, 4,7b, 10b, 13a-hexahidroxytax-11-en 9 one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)- N-benzoyl-3-phenylisoserine.
  Stability: Concentrations of 0.3-1.2 mg/ml in 5% dextrose or normal saline have demonstrated chemical and physical stability for more than 27 hours at ambient temperature (25ºC approximately).
  The intact vial must be stored between 15º and 25ºC.
  Guidelines of Paclitaxel administration: Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  Other Names: Taxol

SUMMARY:
This is an open-label, non-randomised, phase II, multicenter clinical trial. 63 stage IV or stage IIIB/C not candidates for definitive chemo/radiotherapy or surgical resection non-small cell lung cancer (NSCLC) per the 8th edition TNM with no prior systemic anti-cancer therapy will be enrolled in this trial to determine whether therapy decision making based on ctDNA analysis improves overall survival.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, phase II, multicenter clinical trial. The total sample size is 63 patients. The population to be included are stage IV or stage IIIB/C not candidates for definitive chemo/radiotherapy or surgical resection non-small cell lung cancer (NSCLC) per the 8th edition TNM with no prior systemic anti-cancer therap.

Patients will be treated with Cemiplimab for 2 cycles and after response evaluation and ctDNA levels analysis, patients will be treated with Cemiplimab plus chemotherapy or cemiplimab monotherapy depending on response and ctDNA levels.

The primary research goal is to determine whether therapy decision making based on ctDNA analysis improves overall survival.

Patient accrual is expected to be completed within 1.5 years excluding a run-in-period of 4-6 months. An estimated treatment period of 2 years, 2 years of follow-up and the preparation of the final report and the close out visit are expected to extend the study duration to a total of 6.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV or stage IIIB/C not candidates for definitive chemo/radiotherapy or surgical resection non-small cell lung cancer (NSCLC) per the 8th edition TNM with no prior systemic anti-cancer therapy
* PDL1 ≥50%
* ECOG performance status 0-1
* Patients aged ≥ 18 years
* Prior adjuvant or neoadjuvant chemotherapy for early stage is permitted if completed at least 6 months prior to enrolment
* Presence of at least one measurable lesion by CT-scan per RECIST version 1.1
* Anticipated life expectancy >12 weeks
* Correct hematological, hepatic and renal function
* Patient consent must be obtained in the appropriate manner as established in the applicable local and regulatory requirements
* Patients must be accessible for treatment and follow-up
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 3 days before enrolment.
* All sexually active men and women of childbearing potential must use a highly effective contraceptive method during the study treatment and for a period of at least 4 months following the last administration of trial drugs

Exclusion Criteria:

* Patients whose tumors harbor an activating mutation in EGFR, ALK translocation, or ROS Proto-Oncogene 1 (ROS1) rearrangements sensitive to available targeted inhibitor therapy
* Patients with grade ≥2 neuropathy
* Pregnant or breastfeeding women
* Patients with a weight loss >10% within the previous 3 months
* Patients with carcinomatous meningitis
* Patients with a history of other malignant diseases within the past 3 years
* Patients must have recovered from a major surgery at least 14 days prior to enrolment
* Patients with active or uncontrolled infections or with serious medical conditions or disorders that may not allow patient management as established in the protocol
* Prior treatment with antineoplasic drugs or thoracic radiotherapy for any reason different from the ones specific in the inclusion criteria
* Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemo-radiotherapy with curative intent for non-metastatic disease less than 6 months before enrollment since the last chemotherapy, radiotherapy, or chemo-radiotherapy
* Patients with a combination of small cell lung cancer and non-small cell lung cancer, a carcinoid lung tumor or large cell neuroendocrine carcinoma
* Has known allergy or hypersensitivity to components of study drug
* Significant comorbidities that preclude the administration of chemotherapy according to the investigator's criteria
* Ongoing or recent evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments
* Untreated brain metastasis(es) that may be considered active
* Immunosuppressive corticosteroid doses within 4 weeks prior to the first dose of cemiplimab
* Uncontrolled infection with hepatitis B or hepatitis C or human immunodeficiency virus; or diagnosis of immunodeficiency
* History of interstitial lung disease or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management.
* History of documented allergic reactions or acute hypersensitivity reactions attributed to antibody treatments
* Patients with a history of solid organ transplant
* Receipt of live vaccines within 30 days of first study treatment
* Women of childbearing potential, or sexually active men, who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment prior to the start of the first treatment, during the study, and for at least 4 months after the last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2031-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
To determine whether therapy decision making based on ctDNA analysis improves overall survival | From the date of the end of two cycles of Cemiplimab treatment until 24 months
  Test whether the addition of chemotherapy in patients receiving Cemiplimab, based on the ctDNA levels after two cycles of Cemiplimab, improves overall survival (OS) at 24 months. OS defined as the time from enrolment to death from any cause.

SECONDARY OUTCOMES:
To assess the efficacy of the treatment in terms of the Progression Free Survival (PFS) at 12 months | From the date of the end of treatment until 12 months
  PFS defined as the time from enrollment to the first occurrence of disease progression or death from any cause as determined by the investigator according to RECIST v1.1
To evaluate the sites of first failure | From the date of the end of treatment until the date of last follow up, assessed up to 24 months
  To evaluate the sites of first relapse or progression
Duration of response (DOR) | From date of documentation of tumor response until date of first documented progression, assessed up to 24 months
  To evaluate the efficacy of cemiplimab as measured by investigator. Assessed as duration of response (DOR) according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Fundación GECP President
Locations (20):
- Spain (20):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital General de Elche, Elche, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital De Basurto, Bilbao, Bilbao
  - Hospital Universitario Jerez De La Frontera, Jerez de la Frontera, Cádiz
  - Hospital Dr. Josep Trueta, Girona, Girona
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Regional de Málaga, Málaga, Málaga
  - Hospital Universitari Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Universitario Salamanca, Salamanca, Salamanca
  - Hospital General de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org